CLINICAL TRIAL: NCT01190046
Title: Muscle Disuse and Contractile Dysfunction in the Elderly
Brief Title: Chronic Muscle Disuse in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael J. Toth, Ph.D., Associate Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 033547; R01AG033547 (NIH)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Osteoarthritis
Keywords: elderly; muscle; disuse; osteoarthritis; exercise
MeSH Terms: conditions — Osteoarthritis; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resistance exercise training (Other): Exercise is being used as an experimental tool to determine if remediation of muscle disuse counteracts cellular/molecular defects in muscle structure/function.
  Interventions: Behavioral: Resistance exercise training

INTERVENTIONS:
Behavioral: Resistance exercise training — Lower extremity resistance exercise training 3x/wk

SUMMARY:
The purpose of this study is to define the effects of chronic disuse on skeletal muscle structure and function in elderly individuals at the cellular and molecular level by examining elderly characterized by chronic muscle disuse (patients with knee osteoarthritis) and healthy elderly no evidence of knee osteoarthritis and normal physical activity levels.

DETAILED DESCRIPTION:
Skeletal muscle disuse is an important contributing factor to physical disability. Disuse is more frequent in the elderly and they are more susceptible to its debilitating effects because of their diminished physiological reserve. Despite these facts, the mechanisms whereby disuse promotes skeletal muscle contractile dysfunction in this population remain largely undetermined. Therefore, the investigators will systematically test for modifications of single skeletal muscle fiber structure and function that underlie contractile dysfunction. Elderly individuals characterized by chronic muscle disuse (patients with knee osteoarthritis) will be compared to carefully-matched controls with no clinical evidence of knee osteoarthritis and normal activity levels. Thereafter, elderly with chronic disuse will undergo an exercise intervention to remediate muscle disuse. The investigators hypothesize that muscle disuse impairs contractile function, in part, through alterations in myosin kinetics, myofilament protein content and the mechanical properties of the myofilament lattice and that exercise rehabilitation will counteract these deficits. The investigators will specifically examine the effect of disuse on mechanical, kinetic and structural properties and molecular composition of single muscle fibers in cases and controls, as well as determine how increasing muscle use in elderly with chronic disuse via exercise training affects muscle fiber mechanical, kinetic and structural properties and molecular composition. These translational studies will provide the first comprehensive evaluation of the cellular and molecular mechanisms through which muscle disuse alters skeletal muscle structure and contractile function in elderly humans. This knowledge can assist in the development and refinement of preventative and corrective therapies for disability by tailoring these approaches to address specific molecular defects.

ELIGIBILITY:
KNEE OSTEOARTHRITIS PATIENTS

Inclusion Criteria:

* 60-80 yrs of age
* physician-diagnosed, symptomatic knee osteoarthritis
* ambulatory and able to perform lower extremity resistance exercise

Exclusion Criteria:

* rheumatoid arthritis or other autoimmune disease
* chronic heart, lung, kidney or liver disease or hypertension
* diabetes
* history of stroke
* other neurological or musculoskeletal disease

HEALTHY CONTROLS

Criteria are identical to those for knee osteoarthritis patients above, but controls will have no clinical or radiographic evidence of osteoarthritis and will have normal activity physical activity levels.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Single muscle fiber structure/function | Baseline
Single muscle fiber structure/function | 3.5 months (post-training)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Toth, Ph.D., Principal Investigator — University of Vermont and State Agricultural College
Locations (1):
- University of Vermont and State Agricultural College, Burlington, Vermont, United States

REFERENCES:
- [Background] Gustavson AM, Wolfe P, Falvey JR, Eckhoff DG, Toth MJ, Stevens-Lapsley JE. Men and Women Demonstrate Differences in Early Functional Recovery After Total Knee Arthroplasty. Arch Phys Med Rehabil. 2016 Jul;97(7):1154-62. doi: 10.1016/j.apmr.2016.03.007. Epub 2016 Apr 8. PMID 27063363
- [Background] Rengo JL, Callahan DM, Savage PD, Ades PA, Toth MJ. Skeletal muscle ultrastructure and function in statin-tolerant individuals. Muscle Nerve. 2016 Feb;53(2):242-51. doi: 10.1002/mus.24722. Epub 2015 Dec 9. PMID 26059690
- [Background] Miller MS, Bedrin NG, Ades PA, Palmer BM, Toth MJ. Molecular determinants of force production in human skeletal muscle fibers: effects of myosin isoform expression and cross-sectional area. Am J Physiol Cell Physiol. 2015 Mar 15;308(6):C473-84. doi: 10.1152/ajpcell.00158.2014. Epub 2015 Jan 7. PMID 25567808
- [Background] Callahan DM, Bedrin NG, Subramanian M, Berking J, Ades PA, Toth MJ, Miller MS. Age-related structural alterations in human skeletal muscle fibers and mitochondria are sex specific: relationship to single-fiber function. J Appl Physiol (1985). 2014 Jun 15;116(12):1582-92. doi: 10.1152/japplphysiol.01362.2013. Epub 2014 May 1. PMID 24790014
- [Background] Miller MS, Bedrin NG, Callahan DM, Previs MJ, Jennings ME 2nd, Ades PA, Maughan DW, Palmer BM, Toth MJ. Age-related slowing of myosin actin cross-bridge kinetics is sex specific and predicts decrements in whole skeletal muscle performance in humans. J Appl Physiol (1985). 2013 Oct 1;115(7):1004-14. doi: 10.1152/japplphysiol.00563.2013. Epub 2013 Jul 25. PMID 23887900
- [Result] Callahan DM, Tourville TW, Slauterbeck JR, Ades PA, Stevens-Lapsley J, Beynnon BD, Toth MJ. Reduced rate of knee extensor torque development in older adults with knee osteoarthritis is associated with intrinsic muscle contractile deficits. Exp Gerontol. 2015 Dec;72:16-21. doi: 10.1016/j.exger.2015.08.016. Epub 2015 Sep 3. PMID 26343257
- [Result] Callahan DM, Tourville TW, Miller MS, Hackett SB, Sharma H, Cruickshank NC, Slauterbeck JR, Savage PD, Ades PA, Maughan DW, Beynnon BD, Toth MJ. Chronic disuse and skeletal muscle structure in older adults: sex-specific differences and relationships to contractile function. Am J Physiol Cell Physiol. 2015 Jun 1;308(11):C932-43. doi: 10.1152/ajpcell.00014.2015. Epub 2015 Mar 25. PMID 25810256
- [Result] Miller MS, Callahan DM, Toth MJ. Skeletal muscle myofilament adaptations to aging, disease, and disuse and their effects on whole muscle performance in older adult humans. Front Physiol. 2014 Sep 26;5:369. doi: 10.3389/fphys.2014.00369. eCollection 2014. PMID 25309456
- [Result] Callahan DM, Miller MS, Sweeny AP, Tourville TW, Slauterbeck JR, Savage PD, Maugan DW, Ades PA, Beynnon BD, Toth MJ. Muscle disuse alters skeletal muscle contractile function at the molecular and cellular levels in older adult humans in a sex-specific manner. J Physiol. 2014 Oct 15;592(20):4555-73. doi: 10.1113/jphysiol.2014.279034. Epub 2014 Jul 18. PMID 25038243
- [Derived] Voigt TB, Tourville TW, Falcone MJ, Slauterbeck JR, Beynnon BD, Toth MJ. Resistance training-induced gains in knee extensor strength are related to increased neural cell adhesion molecule expression in older adults with knee osteoarthritis. BMC Res Notes. 2019 Sep 18;12(1):595. doi: 10.1186/s13104-019-4642-0. PMID 31533814